CLINICAL TRIAL: NCT05991297
Title: Effects of Deep Sensory Assisted Rehabilitation on Gait and Balance in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nermin Çalışır (Other)
Collaborators: Bursa Sevket Yilmaz Training and Research Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Nermin Çalışır, Principal İnvestigator,Head of Neurology, Romatem Bursa Hospital
Organization: Romatem Bursa Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ROMATEM-NERMİN ÇALIŞIR 2023
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: MS (Multiple Sclerosis)
Keywords: deep sensory assisted rehabilitation; MS gait and balance; deep sensory walkway
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: classic rehabilitation group vs.deep sensory assisted rehabilitation group
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classical physical therapy and rehabilitation program (Active Comparator): Classical rehabilitation program (stretching, strenght, balance and coordination exercise) for fifty minutes.
  Interventions: Other: classical rehabilitation
- Deep sensory asisted therapy and rehabilitation program (Experimental): Deep sensory asisted rehabilitation program (stretching, strenght, balance and coordination and deep sensory exercises) for fifty minutes.
  Interventions: Other: Deep sensory assisted rehabilitation

INTERVENTIONS:
Other: Deep sensory assisted rehabilitation — A new PTR plan called "deep sensory assisted rehabilitation" was created: it was aimed to develop a sensory and deep sense in the adult age group by making use of sensory integration exercises, which are mostly applied in the childhood age group. Whether these exercises are effective on walking and balance will be evaluated. Patients will be dressed in a vest with an equally distributed weight of 4-6 kg according to their weight, and exercises will be done while walking and standing.
  - the so-called "deep sensory pathway"; The patients will be given standing and walking exercises on sand and stone floors, soft floors made of sponge, hard plastic floors with different sizes of grooves and shapes, and hot-cold floors formed by placing hot packs and cold packs.
  Arms: Deep sensory asisted therapy and rehabilitation program
Other: classical rehabilitation — Muscle strengthening in all four extremities; strengthening of trunk and abdominal muscles; providing and maintaining joint range of motion; independent and safe standing, turning, and stepping; able to walk alone on flat ground and on different surfaces (such as sloping-handicapped-soil-stone-sand-grass-rough-stepped)
  Arms: Classical physical therapy and rehabilitation program

SUMMARY:
The effect of physical therapy and rehabilitation on improving the gait and balance disorders of patients has been proven. FTR applications in MS patients have become routine in developed countries. However, due to the high patient density in our country, FTR cannot be performed at the rate we want due to different reasons such as the inability to separate areas special for MS patients, the lack of special FTR applications for MS patients, and the inability to perform regular FTR follow-ups. Even if FTR is recommended and performed, our patients think that FTR is not very effective due to the above reasons and they do not continue.

A team of neurology, physical therapy specialists, and physiotherapists was formed, in-service training was completed and a special rehabilitation program for MS patients was created. First of all, we will apply routine classical FTR to our patients. Sensory and deep sensory disorders, which are more common and severe, especially in the lower extremities, also negatively affect gait and balance.

A rehabilitation program was created by adding exercises to improve sensation and deep sense, along with muscle strengthening. The results of the 1st and 21st sessions of the patients in the two groups who underwent classical rehabilitation and deep sensory-assisted rehabilitation will be compared. It was planned to evaluate the gait and balance parameters of the patients as numerical data with clinical scales and the C mill device we used in walking and balance exercises.

DETAILED DESCRIPTION:
Muscle strengthening in all four extremities; strengthening of trunk and abdominal muscles; providing and maintaining joint range of motion; independent and safe standing, turning, and stepping; able to walk alone on flat ground and on different surfaces (such as sloping-handicapped-soil-stone-sand-grass-rough-stepped); increase in exercise capacity, duration, distance; An increase in the number of steps per minute and step length is expected.

It was thought that both classical rehabilitation and deep sensory-assisted rehabilitation would improve gait and balance parameters.

There has been previous research showing the effects of FTR. What we will do in addition and new with this research;

* The effects of classical rehabilitation and deep sensory-assisted rehabilitation will be compared
* A new PTR plan called "deep sensory assisted rehabilitation" was created: it was aimed to develop a sensory and deep sense in the adult age group by making use of sensory integration exercises, which are mostly applied in the childhood age group. Whether these exercises are effective on walking and balance will be evaluated. Patients will be dressed in a vest with an equally distributed weight of 4-6 kg according to their weight, and exercises will be done while walking and standing.
* the so-called "deep sensory pathway"; The patients will be given standing and walking exercises on sand and stone floors, soft floors made of sponge, hard plastic floors with different sizes of grooves and shapes, and hot-cold floors formed by placing hot packs and cold packs.
* Most of the previous studies have shown the effect of FTR using clinical scales. In developed countries, gait analysis was performed. In our research, we aimed to measure gait and balance parameters in C-mill walking and balance exercise devices, together with clinical scales, as numerical data and graphics. The patient's standing and walking on the treadmill, stride length, stride symmetry, walking speed, distance, duration, cadence, and percentage deviation from targets during tandem and slalom walking parameters will be recorded as objective numerical data and graphics. These measurements will be recorded in the 1st session and the 21st session.

Changes in patients will be seen with clinical scales and visual evaluations. However, in order to make the evaluation more objective for both the patient and the practitioner, these measurements made with the C mill will also be made.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with multiple sclerosis
* 20-60 years old
* EDSS between 3.0-5.5 Those with EDSS 0-2.5 and spinal and/or cerebellar involvement
* Had the last MS attack at least 3 months ago

Exclusion Criteria:

* schizoaffective disorder
* lower extremity amputation
* shortness on one side creating asymmetry in the lower extremities
* diabetes mellitus
* cognitive impairment (at a level that may interfere with communication)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Multipl sclerosis quality of life-54(MSQOL-54) | 1st day: when rehabilitation applications started
  : It is calculated with the combined summary scores of physical and mental health. As the total score increases, the quality of life is evaluated positively.
Multipl sclerosis quality of life-54(MSQOL-54) | after 7 weeks: when rehabilitation applications ended
  : It is calculated with the combined summary scores of physical and mental health. As the total score increases, the quality of life is evaluated positively. The scale has not minimum and maximum value. The change between the participant's prior and values was evaluated.
MiniBest test | 1st day: when rehabilitation applications started
  minimum and maximum score: 0-28: high score indicates good functional balance
MiniBest test | after 7 weeks: when rehabilitation applications ended
  minimum and maximum score: 0-28: high score indicates good functional balance
10 meter walking time | 1st day: when rehabilitation applications started
  The patient's walking time of the determined 10-meter distance is measured.
10 meter walking time | after 7 weeks: when rehabilitation applications ended
  The patient's walking time of the determined 10-meter distance is measured.
Nottingham Extended Activities of Daily Living Scale | 1st day: when rehabilitation applications started
  minimum and maximum score: 0-66: high score indicates no restriction in activities of daily living.
Nottingham Extended Activities of Daily Living Scale | after 7 weeks: when rehabilitation applications ended
  minimum and maximum score: 0-66: high score indicates no restriction in activities of daily living.
Functional Ambulation Classification | 1st day: when rehabilitation applications started
  minimum and maximum score :0-5: high score indicates that walking can be done independently.
Functional Ambulation Classification | after 7 weeks: when rehabilitation applications ended
  minimum and maximum score :0-5: high score indicates that walking can be done independently.
Fatigue Severity Score | 1st day: when rehabilitation applications started
  A score lower than 2.8 indicates no fatigue, a score higher than 6.1 indicates chronic fatigue
Fatigue Severity Score | after 7 weeks: when rehabilitation applications ended
  A score lower than 2.8 indicates no fatigue, a score higher than 6.1 indicates chronic fatigue
DN4(Douleur Neuropathique 4 Questions) | 1st day: when rehabilitation applications started
  Minimum and maximum score: 0-10: A score of 4 and above indicates neuropathic pain.
DN4(Douleur Neuropathique 4 Questions) | after 7 weeks: when rehabilitation applications ended
  Minimum and maximum score: 0-10: A score of 4 and above indicates neuropathic pain.
MSWS-12( MS walking scale-12) | 1st day: when rehabilitation applications started
  minimum and maximum scores: 12-54: low scores indicate that gait disturbance has little effect on disability.
MSWS-12( MS walking scale-12) | after 7 weeks: when rehabilitation applications ended
  minimum and maximum scores: 12-54: low scores indicate that gait disturbance has little effect on disability.
FES-1: (Falls Efficay Scale-1) | 1st day: when rehabilitation applications started
  minimum and maximum score: 16-64: higher score indicates increased anxiety about falling
FES-1: (Falls Efficay Scale-1) | after 7 weeks: when rehabilitation applications ended
  minimum and maximum score: 16-64: higher score indicates increased anxiety about falling

CONTACTS AND LOCATIONS:
Overall Officials: NERMİN ÇALIŞIR, Study Chair — ROMATEM PHYSICAL THERAPY AND REHABILITATION HOSPITALS BURSA HOSPITAL; NURTEN KÜÇÜKÇAKIR, Study Director — ROMATEM PHYSICAL THERAPY AND REHABILITATION HOSPITALS BURSA HOSPITAL; MERAL SEFEROĞLU, Study Director — Bursa Yuksek Ihtisas Training and Research Hospital; ALİ ÖZHAN SIVACI, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital; CELAL BATUHAN GÜNEYSU, Principal Investigator — ROMATEM PHYSICAL THERAPY AND REHABILITATION HOSPITALS BURSA HOSPITAL; İSMAİL HACIOĞLU, Principal Investigator — ROMATEM PHYSICAL THERAPY AND REHABILITATION HOSPITALS BURSA HOSPITAL; YUSUF ZİYA ŞAHİN, Principal Investigator — ROMATEM PHYSICAL THERAPY AND REHABILITATION HOSPITALS BURSA HOSPITAL; MUHAMMED SOC HASANOĞLU, Principal Investigator — ROMATEM PHYSICAL THERAPY AND REHABILITATION HOSPITALS BURSA HOSPITAL; MAHMUT CAN ERDOĞAN, Principal Investigator — ROMATEM PHYSICAL THERAPY AND REHABILITATION HOSPITALS BURSA HOSPITAL; SİNAN ATİLLA, Principal Investigator — ROMATEM PHYSICAL THERAPY AND REHABILITATION HOSPITALS BURSA HOSPITAL
Locations (2):
- Turkey (Türkiye) (2):
  - University of Health Sciences Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Yildirim
  - Romatem Physical Therapy and Rehabilitation Hospitals Bursa Hospital, Bursa